CLINICAL TRIAL: NCT04008862
Title: Characteristics and Effectiveness of a Partnership-based Nursing Practice for Patients With Chronic Lung Diseases and Their Families
Brief Title: Partnership-based Nursing Practice for Lung Patients and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helga Jónsdóttir (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor-Investigator, Helga Jónsdóttir, Professor and Academic Chair of Nursing Care for Chronically Ill Adults, Landspitali University Hospital
Organization: Landspitali University Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: LSH-19-001
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Family; Chronic Disease
Keywords: Chronic Obstructive Pulmonary Disease; Self-management; Palliative care; Family; Chronic Disease; Nursing practice
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Longitudinal design, participants serve as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partnership-based care (Experimental): Each patient will serve as his/her own control
  Interventions: Behavioral: Partnership-based nursing practice

INTERVENTIONS:
Behavioral: Partnership-based nursing practice — Provided by clinical nurse specialists (n=2) and specialized nurses (n=3): i) Partnership-based theoretical nursing practice framework: Family involvement, living with symptoms and access to healthcare -primary goal of enhancement of the health experience. Key question: What are your main concerns about the health of the person with the lung disease? Followed by conversations: a) Existence of lung disease and symptoms that the patient has. b) Nature of disease, its management, quitting smoking, use of inhaler medications, utilization of health care, negative feelings and issues. Skills and motivation to undertake activities to maintain and improve well-being, skills in communication with family, relatives and health professionals. ii) Empirical knowledge about the nature of COPD, symptom management and palliative care and the GOLD clinical guidelines. iii) Patients are seen over an undefined time period in the out-patient clinic or at home depending on needs and capabilities.

SUMMARY:
This study aims to describe and measure the effectiveness of partnership-based nursing care for people with Chronic Obstructive Pulmonary Disease (COPD) and their families. Investigators hypothesize that an holistic, inclusive -taking account of the challenge of multi-morbidity and the long-term relationship that patients with COPD and their families have with the nurses along with the open structure of whatever kind of services is needed in each patient-family case, often in interdisciplinary and inter-institutional collaboration- , is beneficial as regards use of healthcare, health characteristics, HRQL, use of inhaler medications, sense of security in care and illness intrusiveness.

DETAILED DESCRIPTION:
Growing number of people with chronic lung diseases, particularly chronic obstructive pulmonary disease (COPD), and the wide ranging burden that the disease induces to individuals, families and societies, has spurred concerted efforts to develop new healthcare for these people. Outpatient clinics are receiving increasing recognition, particularly those managed by nurses. An out-patient nursing clinic based on theoretical premises of partnership as practice has been established at Landspitali University Hospital. Initial research has shown effectiveness of the practice on the use of healthcare, health status, health related quality of life as well as increased capacity of families to live a meaningful life with the disease. There is a need to substantiate knowledge of the effectiveness of the partnership-based practice by focusing on use of healthcare resources, health and the experience of patients and families, as well as developing educational material for nurses.

Investigators hypothesize that the holistic, inclusive -taking account of the challenge of multi-morbidity and the long-term relationship that patients with COPD and their families have with the nurses along with the open structure of whatever kind of services is needed in each patient-family case, often in interdisciplinary and inter-institutional collaboration- , is beneficial as regards use of healthcare, health characteristics, HRQL, use of inhaler medications, sense of security in care and illness intrusiveness. The experience of patients with COPD and their families of living with the disease and receiving the care will substantiate the previously indicated variables. To this study a multi-dimensional approach is needed which includes both a holistic evaluation (qualitatively studying the experience of participants) and which measures variables prevalent in studies on self-management and palliative care (quantitative use of instruments and demographic variables).

ELIGIBILITY:
Inclusion Criteria:

* Clinical ICD 10 diagnosis of J40 to J44 and J96
* Currently receiving the partnership-based nursing care

Exclusion Criteria:

• Not speaking Icelandic

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life: St. Georges Respiratory Questionnaire 40 item | 18 months
  40 items with Likert-type and dichotomous questions, which are aggregated into a total score and three subscales; symptoms, activity and impacts. Each of the three subscales and the total score is scaled separately in the range 0-100. Higher scores reflect less quality of life. A score change of four units is considered clinically significant.
Hospital Admissions | 18 months
  Numerical scale with frequency from 0 to unknown number

SECONDARY OUTCOMES:
Length of hospital stay | 18 months
  Numerical scale fwith numbers from 0 to unknown number
Hospital Anxiety and Depression Scale | 18 months
  14-item, four-point (0-3) Likert scale with two subscales, anxiety (0-21) and depression (0-21). A mean is calculated for each scale. Higher scores indicates worse condition.
Capacity to use inhalers | 18 months
  Numerical scale 10 item, 4-point Likert type data collection tool. It is has two scales, capacity to inhale medications (5 items) and technical skills to use the inhalers (5 items). Each scale ranges from 0 to 20. A mean is calculated for each score. Higher score indicates better skills in using the inhaler.

OTHER OUTCOMES:
COPD Assessment Test (CAT) | 18 months
  8 items Likert scale (0-5) range from 0 to 40 higher scores indicate lower HRQL.
Modified British Medical Research Council Dyspnea Scale (mMRC) | 18 months
  It is a one item 5-point scale (0-4) based on degrees of various physical activities that precipitate dyspnea. Less dyspnea is indicated by a lower score.
Illness Intrusiveness Rating Scale | 18 months
  IIRS is a 13-item self-reported questionnaire with three subscales, relationships and personal development (passive recreation, family relations, other social relations, self-expression, religious expression and community and civic involvement), intimacy (relationship with your spouse, and sex life) and instrumental (health, work, active recreation and financial situation). One item, diet, is not linked to any of the subscales. A total score is calculated by summing the ratings of all of the items (13-91) and a mean is calculated for each subscale (1-7). Higher score indicates worse outcome.
Sense of Security in Care -Patients' Evaluation (SEC-P) | 18 months
  Items are scored on a six point Likert scale with means calculated for the total scale as well as the 3 subscales: Care (8 item, range 8 to 48), Identity (4 item, range 4 to 32) and Mastery (3 item, range 3 to 24). Higher scores indicate a better outcome. Psychometric properties will be tested in the research.

CONTACTS AND LOCATIONS:
Overall Officials: Helga Jónsdóttir, Principal Investigator — Landspitali. National Hospital of Iceland
Locations (1):
- Landspitali National University Hospital, Reykjavik, Ísland, Iceland

IPD SHARING:
Plan to Share IPD: No